CLINICAL TRIAL: NCT01937663
Title: A Single-blind, Dose-tapering Study of KWA-0711 in Patients With Chronic Constipation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: KWA1203
Record Dates: First submitted 2013-08-27; First posted 2013-09-09 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Chronic Constipation
Keywords: Chronic Constipation; Constipation; Functional gastrointestinal disorders
MeSH Terms: conditions — Constipation; Gastrointestinal Diseases

ARMS (4):
- KWA-0711 Dose1 (Experimental)
  Interventions: Drug: KWA-0711
- KWA-0711 Dose2 (Experimental)
  Interventions: Drug: KWA-0711
- KWA-0711 Dose3 (Experimental)
  Interventions: Drug: KWA-0711
- KWA-0711 Dose4 (Experimental)
  Interventions: Drug: KWA-0711

INTERVENTIONS:
Drug: KWA-0711

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of tapered KWA-0711 dose in chronic constipation patients.

ELIGIBILITY:
Inclusion Criteria:

* The patients who experienced fewer than three spontaneous bowel movements per week for more than 6 months prior to the enrollment.
* The patients who experienced one or more of the following signs or symptoms during more than 25% of bowel movements for more than 6 months: straining, lumpy or hard stools, and a sensation of incomplete evacuation

Exclusion Criteria:

* Patients who have secondary constipation caused by systemic disorder.
* Patients who have organic constipation.
* Patients who received intestinal resection.

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Primary Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Improvement of signs and symptoms associated with constipation | 4 weeks
  * Frequency of Spontaneous Bowel Movements
  * Bowel Movement Timing
  * Stool Consistency
  * Abdominal Assessment
  * QOL Assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Tokyo, Japan